CLINICAL TRIAL: NCT04599413
Title: Transversal Observational Study on Musculoskeletal Disorders in Spanish Pianist
Brief Title: Study on Musculoskeletal Disorders in Spanish Pianist
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Collaborators: ZACARÍAS SANCHEZ MILÁ (Unknown); ANA MARTIN JIMENEZ (Unknown); ANGELICA CAMPON CHEKROUN (Unknown)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, PhD Physiotherapy, Universidad Católica de Ávila
Other Study IDs: 13/10/2020
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Musculoskeletal Diseases
Keywords: assessments; pain; physical therapy specialty; musics
MeSH Terms: conditions — Musculoskeletal Diseases; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SURVEY — Pain survey on pianists

SUMMARY:
Background: musculoskeletal disorders related to instrumental practice (TMRPI) affect many pianists.

Objectives: to know the prevalence of TMRPI in the population of Spanish pianists and its relationship with gender, age, physical activity, number of years playing the piano and the number of hours per week.

Design: transversal study based on a survey that included 30 volunteers of both genders, aged between 17 and 65, who played the piano for at least 2 years.

Method. due to the absence of specific questionnaires for pianist populations on MMRPI, a questionnaire was conducted combining a validated questionnaire on MMR, the Nordic Musculoskeletal Questionnaire (NMQ) with an "ad hoc" questionnaire created specifically for this study

ELIGIBILITY:
Inclusion Criteria:

* over 16 years old
* at least 2 years playing piano

Exclusion Criteria:

* Traumatism

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: professional pianists with musculoskeletal disorders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Pain assessed by VAS Scale | 2 months
  Pain assessed by VAS Scale

SECONDARY OUTCOMES:
YEARS | 2 years
  Incidence of pain over years of practice

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ling CY, Loo FC, Hamedon TR. Playing-Related Musculoskeletal Disorders Among Classical Piano Students at Tertiary Institutions in Malaysia: Proportion and Associated Risk Factors. Med Probl Perform Art. 2018 Jun;33(2):82-89. doi: 10.21091/mppa.2018.2013. PMID 29868681
- [Result] Bragge P, Bialocerkowski A, McMeeken J. A systematic review of prevalence and risk factors associated with playing-related musculoskeletal disorders in pianists. Occup Med (Lond). 2006 Jan;56(1):28-38. doi: 10.1093/occmed/kqi177. Epub 2005 Nov 7. PMID 16275655
- [Result] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Result] Yoshie M, Kudo K, Murakoshi T, Ohtsuki T. Music performance anxiety in skilled pianists: effects of social-evaluative performance situation on subjective, autonomic, and electromyographic reactions. Exp Brain Res. 2009 Nov;199(2):117-26. doi: 10.1007/s00221-009-1979-y. Epub 2009 Aug 22. PMID 19701628
- [Result] Ling CY, Loo FC, Hamedon TR. Knowledge of Playing-Related Musculoskeletal Disorders Among Classical Piano Students at Tertiary Institutions in Malaysia. Med Probl Perform Art. 2016 Dec;31(4):201-204. doi: 10.21091/mppa.2016.4036. PMID 27942698
- [Result] Bruno S, Lorusso A, L'Abbate N. Playing-related disabling musculoskeletal disorders in young and adult classical piano students. Int Arch Occup Environ Health. 2008 Jul;81(7):855-60. doi: 10.1007/s00420-007-0279-8. Epub 2008 Jan 22. PMID 18210148
- [Result] Honarmand K, Minaskanian R, Maboudi SE, Oskouei AE. Electrophysiological assessment of piano players' back extensor muscles on a regular piano bench and chair with back rest. J Phys Ther Sci. 2018 Jan;30(1):67-72. doi: 10.1589/jpts.30.67. Epub 2018 Jan 27. PMID 29410569